CLINICAL TRIAL: NCT06356194
Title: A Phase 1, Open-Label, Multiple Dose Study to Evaluate the Drug-Drug Interaction Potential Between Bemnifosbuvir/Ruzasvir and Bictegravir/Emtricitabine/Tenofovir Alafenamide (Biktarvy®) in Healthy Adult Subjects
Brief Title: Drug-drug Interaction Study of Biktarvy and Bemnifosbuvir/Ruzasvir
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Atea Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: AT-01B-006
Record Dates: First submitted 2024-04-04; First posted 2024-04-10 (Actual); Last update posted 2024-07-31 (Actual); Status verified 2024-07

CONDITIONS: Healthy Volunteer Study
MeSH Terms: interventions — bictegravir, emtricitabine, tenofovir alafenamide, drug combination

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- BEM/RZR vs BEM/RZR + BIK vs BIK (Experimental): n=14
  Interventions: Drug: Cohort 1: Days 1-7 Bemnifosbuvir (BEM)/Ruzasvir (RZR) co-administered. Days 8-17 Bemnifosbuvir (BEM)/Ruzasvir (RZR) co-administered + Biktarvy (BIK). Days 18-24 BIK
- BIK vs BEM/RZR + BIK vs BEM/RZR (Experimental): n=14
  Interventions: Drug: Cohort 2: Days 1-10 Biktarvy (BIK). Days 11-17 Bemnifosbuvir (BEM)/Ruzasvir (RZR) co-administered + Biktarvy (BIK). Days 18-24 Bemnifosbuvir (BEM)/Ruzasvir (RZR) co-administered.

INTERVENTIONS:
Drug: Cohort 1: Days 1-7 Bemnifosbuvir (BEM)/Ruzasvir (RZR) co-administered. Days 8-17 Bemnifosbuvir (BEM)/Ruzasvir (RZR) co-administered + Biktarvy (BIK). Days 18-24 BIK — A co-administered dose of Bemnifosbuvir (BEM)/Ruzasvir (RZR) as separate formulations and Biktarvy (BIK)
  Arms: BEM/RZR vs BEM/RZR + BIK vs BIK
Drug: Cohort 2: Days 1-10 Biktarvy (BIK). Days 11-17 Bemnifosbuvir (BEM)/Ruzasvir (RZR) co-administered + Biktarvy (BIK). Days 18-24 Bemnifosbuvir (BEM)/Ruzasvir (RZR) co-administered. — A co-administered dose of Bemnifosbuvir (BEM)/Ruzasvir (RZR) as separate formulations and Biktarvy (BIK)
  Arms: BIK vs BEM/RZR + BIK vs BEM/RZR

SUMMARY:
Drug-drug interaction study of Biktarvy and Bemnifosbuvir/Ruzasvir

ELIGIBILITY:
Inclusion Criteria:

* Must agree to use two methods of birth control from Screening through 90 days after administration of the last dose of study drug.
* Minimum body weight of 50 kg and body mass index (BMI) of 18-30 kg/m2.
* Willing to comply with the study requirements and to provide written informed consent.

Exclusion Criteria:

* Infected with hepatitis B virus, hepatitis C virus, HIV or SARS-CoV-2.
* Abuse of alcohol or drugs.
* Use of other investigational drugs within 28 days of dosing.
* Concomitant use of prescription medications, or systemic over-the-counter medications.
* Other clinically significant medical conditions or laboratory abnormalities.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 28 (Actual)
Dates: Start 2024-04-15 (Actual); Primary Completion 2024-05-30 (Actual); Study Completion 2024-05-30 (Actual)

PRIMARY OUTCOMES:
PK of Biktarvy (BIK: Bictegravir, tenofovir alafenamide, emtricitabine) on the pharmacokinetics (PK) of Bemnifosbuvir (BEM) and Ruzasvir (RZR). | Day 2, Days 4-7, Days 14-17, Days 21-24
  Maximum plasma concentration (Cmax) and Area under the plasma concentration-time curve (AUC)
To determine the effect of Bemnifosbuvir (BEM)/Ruzasvir (RZR) combination on the PK of Biktarvy (BIK: Bictegravir, tenofovir alafenamide, emtricitabine) | Days 7-10, Day 12, Days 14-17, Days 21-24.
  Maximum plasma concentration (Cmax) and Area under the plasma concentration-time curve (AUC)

CONTACTS AND LOCATIONS:
Locations (1):
- Atea Study Site, Québec, Montreal, Canada

IPD SHARING:
Plan to Share IPD: No